CLINICAL TRIAL: NCT05381077
Title: Evaluation of Whole Body Examination by MRI Integrating the "Zero Time Eco" Sequence (ZTE, Pseudo-CT) for the Detection of Bone Lesions in Multiple Myeloma: Comparison With Pet / CT and Whole Body Scanner
Acronym: MM-ZTE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Lecouvet, Prof, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020/27JUL/380
Record Dates: First submitted 2022-05-04; First posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Multiple Myeloma; Bone Metastases
Keywords: MRI; Zero time echo
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: Whole body MRI in addition to the classic PET / CT assessment for all participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Whole body MRI (Other): There is only one cohort where each patient have the standard of care follow up (PET/CT) and Whole body MRI- ZTE sequence for the study
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — Whole body MRI (ZTE sequence)

SUMMARY:
To assess the added value of magnetic resonance imaging (MRI) of the skeleton compared to other validated techniques for the detection of bone lesions in patients with multiple myeloma.

DETAILED DESCRIPTION:
The aim of our study is to offer patients benefiting from a diagnostic approach to myeloma by PET / CT, a whole body MRI examination (MRI-CE) comprising, in addition to the "classic bone marrow" sequences, a ZTE sequence (see below) . This study is being undertaken to compare and assess the complementarity of imaging techniques in the diagnostic management of this disease.

The stages of the work will be:

Optimizing bone marrow exploration sequences by MRI (F. Lecouvet, N. Michoux, Gaetan Duchêne).

Develop and validate a whole body-wide new MRI sequence "ZTE" capable of detecting and quantifying disease-induced osteolysis in the skeleton.

Optimize the reconstruction of these images (Deep Learning software developed with the firm GE), training of the reconstruction of ZTE images by correlation with the scanner (F. Lecouvet, N. Michoux, Gaetan Duchêne).

This approach is completely original, never having been evaluated: the ZTE sequence is a recent development, made available at CUSL on the new research MRI magnet.

The addition of this sequence to the already major information provided by MRI for the detection of the disease and the evaluation of its response (method of choice, see below) would constitute a major advance in establishing the diagnostic value of this technique. non-irradiating compared to other techniques (PET-CT, low dose scanner, etc.).

ELIGIBILITY:
Inclusion Criteria:

* Patient with newly diagnosed multiple myeloma, for whom bone imaging is required for staging.
* Recurrent patient after intensive treatment (high dose chemotherapy, bone marrow transplant, etc.).
* Patient requiring a PET / CT considered as the technique of choice in these stages of the disease.

Exclusion Criteria:

* Implanted material incompatible with MRI.
* Severe claustrophobia.
* Pregnant women

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-02-02 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the diagnostic performance of the different imaging protocols | through study completion, an average of 1 year
  The diagnostic performance of the different imaging protocols will be evaluated by analyzing the receptor efficiency function (ROC curve) and by estimating the Sensitivity (Se), Specificity (Sp), Positive Predictive Value (PPV), Negative Predictive Value (NPV) ) as well as the Predictive Accuracy (Acc) of the different imaging protocols.
Comparison of Sensitivity (Se) and Predictive Precision (Acc) of the different imaging protocols | through study completion, an average of 1 year
  McNemar test on paired data. The Gold Standard will be determined by a panel of independent experts based on all available imaging techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Frederic Lecouvet, MD-PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques Universaires Siant Luc, Brussels, Belgium

REFERENCES:
- [Derived] Chabot C, Haegeman M, Chaouch E, Dumitriu D, Menten R, Steenhaut P, Bernard P, Triqueneaux P, Michoux N, Lecouvet FE. MRI-based pseudo-CT sequences as a radiation-free alternative to CT for obstetric pelvimetry: a proof-of-concept study. Eur Radiol Exp. 2025 May 19;9(1):52. doi: 10.1186/s41747-025-00585-y. PMID 40388042
- [Derived] Lecouvet FE, Zan D, Lepot D, Chabot C, Vekemans MC, Duchene G, Chiabai O, Triqueneaux P, Kirchgesner T, Taihi L, Poujol J, Gheysens O, Michoux N. MRI-based Zero Echo Time and Black Bone Pseudo-CT Compared with Whole-Body CT to Detect Osteolytic Lesions in Multiple Myeloma. Radiology. 2024 Oct;313(1):e231817. doi: 10.1148/radiol.231817. PMID 39377681